CLINICAL TRIAL: NCT01634165
Title: Pharmacokinetics and Pharmacodynamics of LY2963016 Compared to Lantus® in Healthy Subjects Following Two Single Subcutaneous Doses
Brief Title: A Study of LY2963016 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 14676; I4L-MC-ABEM (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-07-02; First posted 2012-07-06 (Estimated); Results first posted 2014-10-07 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — LY2963016 insulin glargine; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0.3 U/kg LY2963016 (Experimental): Single 0.3 units/kilogram (U/kg) subcutaneous dose of LY2963016
  Interventions: Drug: LY2963016
- 0.3 U/kg Lantus (Experimental): Single 0.3 U/kg subcutaneous dose of Lantus
  Interventions: Drug: Lantus
- 0.6 U/kg LY2963016 (Experimental): Single 0.6 U/kg subcutaneous dose of LY2963016
  Interventions: Drug: LY2963016
- 0.6 U/kg Lantus (Experimental): Single 0.6 U/kg subcutaneous dose of Lantus
  Interventions: Drug: Lantus

INTERVENTIONS:
Drug: LY2963016 — Administered subcutaneously
  Arms: 0.3 U/kg LY2963016; 0.6 U/kg LY2963016
Drug: Lantus — Administered subcutaneously
  Arms: 0.3 U/kg Lantus; 0.6 U/kg Lantus

SUMMARY:
This study involves 2 single injections of LY2963016 and 2 single injections of Lantus. There will be at least 6 days between each injection.

The study will compare LY2963016 to Lantus at two different doses.

This study is approximately 10 weeks long, not including screening. Screening is required within 4 weeks of the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females
* Women must be either surgically sterile, post-menopausal, or agree to use a reliable method of birth control during the study
* Have a body mass index between 18.5 and 29.9 kilograms per meter squared (kg/m²)
* Are nonsmokers and have not smoked for at least 6 months prior to entering the study
* Have normal blood pressures and pulse rates at screening, as determined by the investigator
* Have an electrocardiogram (ECG) at screening considered as within normal limits by the investigator
* Have clinical laboratory test results within normal reference range for the population
* Have fasting plasma glucose <110 milligrams per deciliter (mg/dL) (<6.0 micromoles per liter [mmol/L]) at screening
* Have venous access sufficient to allow for blood sampling, intravenous drug administration, and clamp procedures as per the protocol
* Have given written informed consent approved by Lilly and the ethical review board (ERB) governing the site

Exclusion Criteria:

* Are persons who have previously completed or withdrawn from this study
* Are currently enrolled in or have discontinued within the last 30 days from a clinical trial involving an investigational drug or device or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin
* Have significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Show evidence of significant active neuropsychiatric disease
* Show evidence of current use of known drugs of abuse or have a history of use within the past year
* Have a history of first-degree relatives known to have diabetes mellitus
* Show evidence of an acute infection with fever or infectious disease at the time of study entry
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies at screening
* Have positive hepatitis B surface antigens at screening
* Intend to use over-the-counter medication within 7 days or prescription medication within 14 days prior to dosing (apart from vitamin/mineral supplements, occasional paracetamol, thyroid replacement, or birth control methods)
* Have donated blood or had a blood loss of 450 milliliters (mL) 3 months prior to study enrollment
* Have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females) or are unwilling to stop alcohol consumption from 48 hours prior to each dosing until discharged from the clinical research unit (CRU)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a 4-treatment, 4-period, crossover, euglycemic clamp study. Participants were randomly assigned to 1 of 4 dosing sequences.
Groups:
- 0.3 U/kg LY, 0.6 U/kg LY, 0.3 U/kg Lantus, 0.6 U/kg Lantus: Single subcutaneous dose of 0.3 units/kilogram (U/kg) LY2963016 during Period 1; Single subcutaneous dose of 0.6 U/kg LY2963016 during Period 2; Single subcutaneous dose of 0.3 U/kg Lantus during Period 3; Single subcutaneous dose of 0.6 U/kg Lantus during Period 4. There was a minimum washout interval of 6 days between each period.
- 0.6 U/kg LY, 0.6 U/kg Lantus, 0.3 U/kg LY, 0.3 U/kg Lantus: Single subcutaneous dose of 0.6 U/kg LY2963016 during Period 1; Single subcutaneous dose of 0.6 U/kg Lantus during Period 2; Single subcutaneous dose of 0.3 U/kg LY2963016 during Period 3; Single subcutaneous dose of 0.3 U/kg Lantus during Period 4. There was a minimum washout interval of 6 days between each period.
- 0.3 U/kg Lantus, 0.3 U/kg LY, 0.6 U/kg Lantus, 0.6 U/kg LY: Single subcutaneous dose of 0.3 U/kg Lantus during Period 1; Single subcutaneous dose of 0.3 U/kg LY2963016 during Period 2; Single subcutaneous dose of 0.6 U/kg Lantus during Period 3; Single subcutaneous dose of 0.6 U/kg LY2963016 during Period 4. There was a minimum washout interval of 6 days between each period.
- 0.6 U/kg Lantus, 0.3 U/kg Lantus, 0.6 U/kg LY, 0.3 U/kg LY: Single subcutaneous dose of 0.6 U/kg Lantus during Period 1; Single subcutaneous dose of 0.3 U/kg Lantus during Period 2; Single subcutaneous dose of 0.6 U/kg LY2963016 during Period 3; Single subcutaneous dose of 0.3 U/kg LY2963016 during Period 4. There was a minimum washout interval of 6 days between each period.
Period: Period 1
Arm/Group | 0.3 U/kg LY, 0.6 U/kg LY, 0.3 U/kg Lantus, 0.6 U/kg Lantus | 0.6 U/kg LY, 0.6 U/kg Lantus, 0.3 U/kg LY, 0.3 U/kg Lantus | 0.3 U/kg Lantus, 0.3 U/kg LY, 0.6 U/kg Lantus, 0.6 U/kg LY | 0.6 U/kg Lantus, 0.3 U/kg Lantus, 0.6 U/kg LY, 0.3 U/kg LY
Started | 6 | 6 | 6 | 6
Received at Least 1 Dose of Study Drug | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | 0.3 U/kg LY, 0.6 U/kg LY, 0.3 U/kg Lantus, 0.6 U/kg Lantus | 0.6 U/kg LY, 0.6 U/kg Lantus, 0.3 U/kg LY, 0.3 U/kg Lantus | 0.3 U/kg Lantus, 0.3 U/kg LY, 0.6 U/kg Lantus, 0.6 U/kg LY | 0.6 U/kg Lantus, 0.3 U/kg Lantus, 0.6 U/kg LY, 0.3 U/kg LY
Started | 6 | 6 | 6 | 6
Completed | 6 | 5 | 6 | 6
Not Completed | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Period: Period 3
Arm/Group | 0.3 U/kg LY, 0.6 U/kg LY, 0.3 U/kg Lantus, 0.6 U/kg Lantus | 0.6 U/kg LY, 0.6 U/kg Lantus, 0.3 U/kg LY, 0.3 U/kg Lantus | 0.3 U/kg Lantus, 0.3 U/kg LY, 0.6 U/kg Lantus, 0.6 U/kg LY | 0.6 U/kg Lantus, 0.3 U/kg Lantus, 0.6 U/kg LY, 0.3 U/kg LY
Started | 6 | 5 | 6 | 6
Completed | 6 | 5 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | 0.3 U/kg LY, 0.6 U/kg LY, 0.3 U/kg Lantus, 0.6 U/kg Lantus | 0.6 U/kg LY, 0.6 U/kg Lantus, 0.3 U/kg LY, 0.3 U/kg Lantus | 0.3 U/kg Lantus, 0.3 U/kg LY, 0.6 U/kg Lantus, 0.6 U/kg LY | 0.6 U/kg Lantus, 0.3 U/kg Lantus, 0.6 U/kg LY, 0.3 U/kg LY
Started | 6 | 5 | 6 | 6
Completed | 6 | 5 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who received at least one dose of study drug.
Groups:
- All Participants: Single subcutaneous dose of 0.3 units/kilogram (U/kg) LY2963016, or 0.6 U/kg LY2963016, or 0.3 U/kg Lantus, or 0.6 U/kg Lantus during 1 of the 4 study periods in 1 of the 4 study sequences. There was a minimum washout interval of 6 days between each period.
Arm/Group | All Participants
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.1 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 20
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 24
Region of Enrollment [Number; unit: participants]
  Singapore | 24

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Serum LY2963016 or Lantus Concentration-Time Curve (AUC) From Zero to Infinity [AUC(0-∞)]
Description: Results for LY2936016 treatment arms provide the AUC(0-∞) data for LY2936016, while the results for Lantus treatment arms provide the AUC(0-∞) for Lantus.
Time Frame: Predose up to 24 hours after administration of study drug
Population: All participants who received study drug and had sufficient pharmacokinetic data to calculate AUC(0-∞). Participants were analyzed based on the treatment they received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomoles*hour per liter (pmol*h/L)
Groups:
- 0.3 U/kg LY2963016: Single subcutaneous dose of 0.3 units/kilogram (U/kg) LY2963016 during 1 of the 4 study periods in 1 of the 4 study sequences. There was a minimum washout interval of 6 days between each period.
- 0.6 U/kg LY2963016: Single subcutaneous dose of 0.6 U/kg LY2963016 during 1 of the 4 study periods in 1 of the 4 study sequences. There was a minimum washout interval of 6 days between each period.
- 0.3 U/kg Lantus: Single subcutaneous dose of 0.3 U/kg Lantus during 1 of the 4 study periods in 1 of the 4 study sequences. There was a minimum washout interval of 6 days between each period.
- 0.6 U/kg Lantus: Single subcutaneous dose of 0.6 U/kg Lantus during 1 of the 4 study periods in 1 of the 4 study sequences. There was a minimum washout interval of 6 days between each period.
Arm/Group | 0.3 U/kg LY2963016 | 0.6 U/kg LY2963016 | 0.3 U/kg Lantus | 0.6 U/kg Lantus
Number analyzed (Participants) | 23 | 24 | 22 | 24
picomoles*hour per liter (pmol*h/L) | 2330 (39) | 4470 (15) | 2390 (33) | 4310 (51)

2. Primary Outcome: Pharmacokinetics: Maximum Serum LY2963016 or Lantus Concentration (Cmax)
Time Frame: Predose up to 24 hours after administration of study drug
Population: All participants who received study drug and had sufficient pharmacokinetic data to calculate Cmax. Participants were analyzed based on the treatment they received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomoles per liter (pmol/L)
Arm/Group | 0.3 U/kg LY2963016 | 0.6 U/kg LY2963016 | 0.3 U/kg Lantus | 0.6 U/kg Lantus
Number analyzed (Participants) | 23 | 24 | 23 | 24
picomoles per liter (pmol/L) | 108 (20) | 180 (28) | 105 (33) | 174 (38)

3. Secondary Outcome: Pharmacokinetics: Area Under the Serum Concentration-Time Curve From Time Zero to 24 Hours [AUC(0-24)] of LY2963016 or Lantus
Description: Results for LY2936016 treatment arms provide the AUC(0-24) data for LY2936016, while the results for Lantus treatment arms provide the AUC(0-24) for Lantus.
Time Frame: Predose up to 24 hours after administration of study drug
Population: All participants who received study drug and had sufficient pharmacokinetic data to calculate AUC(0-24). Participants were analyzed based on the treatment they received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomoles*hour per liter (pmol*h/L)
Arm/Group | 0.3 U/kg LY2963016 | 0.6 U/kg LY2963016 | 0.3 U/kg Lantus | 0.6 U/kg Lantus
Number analyzed (Participants) | 23 | 24 | 23 | 24
picomoles*hour per liter (pmol*h/L) | 1730 (20) | 3160 (27) | 1690 (30) | 2940 (45)

4. Secondary Outcome: Pharmacokinetics: Area Under the Serum Concentration-Time Curve (AUC) From Time Zero to Last Measured Concentration Value [AUC(0-tlast)] of LY2963016 or Lantus
Description: Results for LY2936016 treatment arms provide the AUC(0-tlast) data for LY2936016, while the results for Lantus treatment arms provide the AUC(0-tlast) for Lantus.
Time Frame: Predose up to 24 hours after administration of study drug
Population: All participants who received study drug and had sufficient pharmacokinetic data to calculate AUC(0-tlast). Participants were analyzed based on the treatment they received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomoles*hour per liter (pmol*h/L)
Arm/Group | 0.3 U/kg LY2963016 | 0.6 U/kg LY2963016 | 0.3 U/kg Lantus | 0.6 U/kg Lantus
Number analyzed (Participants) | 23 | 24 | 23 | 24
picomoles*hour per liter (pmol*h/L) | 1730 (20) | 3160 (27) | 1670 (28) | 2940 (45)

5. Secondary Outcome: Maximum Glucose Infusion Rate (Rmax)
Description: Rmax is used to measure the study drug action over time as measured by the euglycaemic clamp procedure. During the euglycaemic clamp procedure, blood glucose concentrations are held constant after the administration of LY2963016 or Lantus by adjusting the exogenous glucose infusion rate.
Time Frame: Postdose up to 24 hours after administration of study drug
Population: All participants who received study drug and had Rmax measurements. Participants were analyzed based on the treatment they received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams/kilograms/minute (mg/kg/min)
Arm/Group | 0.3 U/kg LY2963016 | 0.6 U/kg LY2963016 | 0.3 U/kg Lantus | 0.6 U/kg Lantus
Number analyzed (Participants) | 23 | 24 | 23 | 24
milligrams/kilograms/minute (mg/kg/min) | 1.81 (100) | 3.05 (59) | 1.70 (92) | 3.25 (54)

6. Secondary Outcome: Total Amount of Glucose Infused (Gtot)
Description: Gtot is used to measure the study drug action over time as measured by the euglycaemic clamp procedure. During the euglycaemic clamp procedure, blood glucose concentrations are held constant after the administration of LY2963016 or Lantus by adjusting the exogenous glucose infusion rate.
Time Frame: Postdose up to 24 hours after administration of study drug
Population: All participants who received study drug and had Gtot measurements. Participants were analyzed based on the treatment they received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams per kilograms (mg/kg)
Arm/Group | 0.3 U/kg LY2963016 | 0.6 U/kg LY2963016 | 0.3 U/kg Lantus | 0.6 U/kg Lantus
Number analyzed (Participants) | 23 | 24 | 23 | 24
milligrams per kilograms (mg/kg) | 1060 (178) | 2260 (80) | 1050 (130) | 2590 (62)

ADVERSE EVENTS:
Arm/Group | 0.3 U/kg LY2963016 | 0.6 U/kg LY2963016 | 0.3 U/kg Lantus | 0.6 U/kg Lantus
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24 | 0/23 | 1/24
Other Adverse Events (participants affected / at risk) | 4/23 | 10/24 | 10/23 | 12/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.3 U/kg LY2963016 (N=23) | 0.6 U/kg LY2963016 (N=24) | 0.3 U/kg Lantus (N=23) | 0.6 U/kg Lantus (N=24)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.3 U/kg LY2963016 (N=23) | 0.6 U/kg LY2963016 (N=24) | 0.3 U/kg Lantus (N=23) | 0.6 U/kg Lantus (N=24)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (3)
Application site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Application site haematoma (General disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural swelling (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 3 (3) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 4 (4) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes